CLINICAL TRIAL: NCT03499054
Title: Breathing Exercises to Improve Fatigue and Quality of Life in Hemodialysis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taipei University of Nursing and Health Sciences (Other)
Responsible Party: Principal Investigator, HUANG HSIN YI, Co-head of Nurses, AHN Department of Internal Medicine, National Taipei University of Nursing and Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 4rfvgy7m
Record Dates: First submitted 2018-01-31; First posted 2018-04-17 (Actual); Last update posted 2018-04-17 (Actual); Status verified 2018-02

CONDITIONS: Hemodialysis; Breathing Exercises; Fatigue
Keywords: Breathing exercises; fatigue; quality of life
MeSH Terms: conditions — Fatigue | interventions — Breathing Exercises

STUDY DESIGN:
Intervention Model Description: Randomized hemodialysis patients in hospital
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (No Intervention): Hemodialysis patients in the control group who receive only routine nursing care during hemodialysis
- exercise group (Experimental): The exercise group are asked to perform breathing exercises during hemodialysis for the study period of 3 months.
  Interventions: Other: Breathing exercises

INTERVENTIONS:
Other: Breathing exercises — During hemodialysis, the participants in the exercise group are asked to keep ttheir muscles relaxed, breathe normally through the nose at a rate of 3-8 times per minute with each breath held over 5 seconds in length. At the same time, the particpants are asked to also perform lower leg lifts for about 8 seconds per lift. The exercise is performed for 15-20 minutes, and after resting, blood pressure, oxygen saturation and HRV are measured.
  Arms: exercise group

SUMMARY:
Breathing exercises to improve fatigue and quality of life in hemodialysis patients

DETAILED DESCRIPTION:
Patients receiving haemodialysis have poor physical function, psychological status and quality of life than the general population.Fatigue is a debilitating symptom in haemodialysis patients Exercise training may improve these parameters for haemodialysis patients.

A 3-month randomized control trial with baseline、Week 4、Week 12 measurement periods was conducted. Exercise group was taught to Breathing exercise week and Usual care for three months. The control group received usual routine care.

A total of 86 patients participated in this study, with 43 patients in the Exercise group and 43 patients in the control group Methods: Hemodialysis Fatigue scale 、 WHOQOL-BREF 、 HADS_ Anxiety

、 HRV

ELIGIBILITY:
Inclusion Criteria:

1. diagnosed by end-stage renal disease, regular hemodialysis three times a week and up to six months or more
2. Adults over 20 years of age.
3. Consciousness.
4. can be used to communicate in Taiwanese, accept questionnaire interviews or self-filling questionnaire.
5. no chest pain or shortness of breath symptoms.
6. No lower extremity disability and ability to walk on their own.
7. agree to take respiratory exercise intervention measures, have the intention to participate in this study and signed a consent form.

Exclusion Criteria:

1. unstable vital signs, or serious heart disease: such as the diagnosis of myocardial infarction, unstable angina pectoris, cardiopulmonary disease and other patients.
2. A complication occurs, such as aspiration pneumonia.
3. history of arrhythmia, as well as taking heart rate medication.
4. Physician's advice is not suitable for exercise, such as bone and joint problems.
5. There is a temporary double vena cava catheter placed.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2017-06-15 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
fatigue | A 3-month
  Assessment of fatigue using fatigue score with a lowest score of 26 points and highest score of 104 points in the control group and the exercise group at the start of the study(baseline), Week 4 and Week 12 for a total of A 3-month

SECONDARY OUTCOMES:
quality of life | A 3-month
  Assessment of quality of life score using WHOQOL-BREF with a lowest score of 26 points and highest score of 130 points in the control group and the exercise group at the start of the study (baseline), Week 4 and Week 12 for a total of A 3-month

CONTACTS AND LOCATIONS:
Locations (1):
- Far Eastern Memorial Hospital, Taipei County, Taiwan

IPD SHARING:
Plan to Share IPD: No